CLINICAL TRIAL: NCT05235685
Title: Impaired Tissue Oxygen Delivery in Patients With Coexistent COPD-heart Failure: What Consequences on Neuromuscular Fatigue During Exercise?
Brief Title: Neuromuscular Fatigue During Exercise in COPD-HF Overlap
Acronym: FIBOX
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021-A02359-32
Record Dates: First submitted 2022-01-18; First posted 2022-02-11 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Heart Failure
Keywords: Exercise Tolerance; Hypoxia, Brain; Muscle Fatigue; Oxygen; Spectroscopy, Near-Infrared; Ultrasonography, Doppler, Transcranial
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Heart Failure; Hypoxia, Brain | interventions — Air

STUDY DESIGN:
Intervention Model Description: 2 parralel study groups: patients with COPD (N=20); patients with COPD-HF overlap (N=20) Between-group comparison (COPD vs COPD-HF) under medical air Only patients with COPD-HF overlap exposed to intervention (hyperoxia)
Who Masked: Participant
Masking Description: Patients masked from intervention (gas mixture being delivered). Non-randomized (air medical condition tested first).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with COPD (Active Comparator): Patients with COPD will only exercise under medical air (for between-group comparison: COPD vs COPD-HF)
  Interventions: Other: Medical air
- Patients with COPD-HF overlap (Experimental): Patients with COPD-HF overlap will first exercise under medical air (for between-group comparison: COPD vs COPD-HF); Patients with COPD-HF overlap will then exercise under intervention (hyperoxia, for within-group comparison: medical air vs intervention trial)
  Interventions: Other: Medical air; Other: Hyperoxia

INTERVENTIONS:
Other: Medical air — Exercise under medical air, both arms exposed.
Other: Hyperoxia — Exercise under hyperoxia, only experimental arm exposed.
  Arms: Patients with COPD-HF overlap

SUMMARY:
Rationale. Chronic obstructive pulmonary disease (COPD) and heart failure (HF) coexist in approximately one third of patients presenting with one of these conditions. From a clinical standpoint, impaired tissue oxygen (O2) delivery stands as a common pathological mechanism of these cardiorespiratory diseases. Recent evidence suggest that muscle and cerebral blood flow and oxygenation are further impaired during exercise in patients with COPD-HF overlap compared to isolated diseases. However, it remains unknown whether impaired O2 delivery is associated with exaggerated manifestations of peripheral and central fatigue in COPD-HF overlap. In addition, improving cardiopulmonary interactions through non invasive positive pressure ventilation or through the addition of a hyperoxic gas mixture during exercise have been associated with enhanced cerebral and muscle O2 delivery and oxygenation in patients with COPD or HF. It is, therefore, conceivable that improved O2 delivery to these structures have beneficial influence on exercise capacity in patients with COPD-HF overlap due to less peripheral and central fatigue.

Aims. To investigate the influence of impaired O2 delivery during exercise, and its alleviation with different interventions (non invasive positive pressure ventilation or hyperoxia), on neuromuscular fatigue in patients with COPD-HF.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* COPD: mild-to-severe airflow obstruction (forced expiratory volume in 1 second (FEV1)/forced vital capacity ratio <0.70; post-bronchodilator FEV1 > 30% predicted);
* HF: reduced left ventricular ejection fraction (<50%, for COPD-HF patients only);
* HF: New York Heart Association Functional Classification I to III (for COPD-HF patients only);
* Clinical stability for both diseases (COPD and/or HF) and no recent (within 3 months) exacerbation requiring a change in medications;
* Patient benefiting from health care coverage;
* Patient able to provide written informed consent.

Exclusion Criteria:

* Inability to perform cycle ergometry;
* Medical device incompatible with magnetic stimulation;
* Counter-indication to perform exercise test;
* Patient refusing to sign written informed consent;
* Patient not benefiting from health care coverage;
* Patient exceeding the annual ceiling of authorized compensation received following participation to a clinical trial;
* Patient deprived of freedom by judicial or administrative decision;
* Patient subject to a measure of legal protection (safeguard of justice, guardianship, curatorship), who cannot be included in clinical trials;
* Pregnant or nursing woman.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-02-21 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Muscle fatigue | Muscle fatigue assessed immediately after exercise, between-group (COPD vs COPD-HF under medical air) and within-group (medical air vs intervention trial in COPD-HF) comparisons
  Muscle fatigue assessed by magnetic stimulation of the femoral nerve

SECONDARY OUTCOMES:
Exertional symptoms | Symptoms during exercise, between-group (COPD vs COPD-HF under medical air) and within-group (medical air vs intervention trial in COPD-HF) comparisons
  Symptoms of dyspnea, leg discomfort, and fatigue
Tissue oxygenation | Tissue oxygenation during exercise, between-group (COPD vs COPD-HF under medical air) and within-group (medical air vs intervention trial in COPD-HF) comparisons
  Prefrontal and quadriceps oxygenation (near-infrared spectroscopy)
Cerebral blood flow | Cerebral blood flow during exercise, between-group (COPD vs COPD-HF under medical air) and within-group (medical air vs intervention trial in COPD-HF) comparisons
  Middle cerebral artery blood flow velocity (transcranial Doppler ultrasonography)
Cardiac output | Cardiac output during exercise, between-group (COPD vs COPD-HF under medical air) and within-group (medical air vs intervention trial in COPD-HF) comparisons
  Cardiac output (signal-morphology impedance cardiography)

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane Doutreleau, MD, PhD, Principal Investigator — CHU Grenoble Alpes, Grenoble Alpes University; Mathieu Marillier, PhD, Study Chair — CHU Grenoble Alpes, Grenoble Alpes University
Locations (1):
- CHU Grenoble Alpes - Hopital Sud (Laboratoire HP2), Échirolles, Auvergne-Rhône-Alpes, France

IPD SHARING:
Plan to Share IPD: Yes
Data will be available on reasonable request to the Investigators (unidentified patients' data).
Time Frame: Data will be available on reasonable request to the Investigators (unidentified patients' data) upon study completion and for an unrestricted period of time.
Access Criteria: Data available on reasonable request to the Investigators.

REFERENCES:
- [Background] Rutten FH, Cramer MJ, Grobbee DE, Sachs AP, Kirkels JH, Lammers JW, Hoes AW. Unrecognized heart failure in elderly patients with stable chronic obstructive pulmonary disease. Eur Heart J. 2005 Sep;26(18):1887-94. doi: 10.1093/eurheartj/ehi291. Epub 2005 Apr 28. PMID 15860516
- [Background] Oliveira MF, Zelt JT, Jones JH, Hirai DM, O'Donnell DE, Verges S, Neder JA. Does impaired O2 delivery during exercise accentuate central and peripheral fatigue in patients with coexistent COPD-CHF? Front Physiol. 2015 Jan 7;5:514. doi: 10.3389/fphys.2014.00514. eCollection 2014. PMID 25610401
- [Background] Oliveira MF, Alencar MC, Arbex F, Souza A, Sperandio P, Medina L, Medeiros WM, Hirai DM, O'Donnell DE, Neder JA. Effects of heart failure on cerebral blood flow in COPD: Rest and exercise. Respir Physiol Neurobiol. 2016 Jan 15;221:41-8. doi: 10.1016/j.resp.2015.10.005. Epub 2015 Oct 31. PMID 26528895
- [Background] Oliveira MF, Arbex FF, Alencar MC, Souza A, Sperandio PA, Medeiros WM, Mazzuco A, Borghi-Silva A, Medina LA, Santos R, Hirai DM, Mancuso F, Almeida D, O'Donnell DE, Neder JA. Heart Failure Impairs Muscle Blood Flow and Endurance Exercise Tolerance in COPD. COPD. 2016 Aug;13(4):407-15. doi: 10.3109/15412555.2015.1117435. Epub 2016 Jan 20. PMID 26790095
- [Background] Borghi-Silva A, Oliveira CC, Carrascosa C, Maia J, Berton DC, Queiroga F Jr, Ferreira EM, Almeida DR, Nery LE, Neder JA. Respiratory muscle unloading improves leg muscle oxygenation during exercise in patients with COPD. Thorax. 2008 Oct;63(10):910-5. doi: 10.1136/thx.2007.090167. Epub 2008 May 20. PMID 18492743
- [Background] Borghi-Silva A, Carrascosa C, Oliveira CC, Barroco AC, Berton DC, Vilaca D, Lira-Filho EB, Ribeiro D, Nery LE, Neder JA. Effects of respiratory muscle unloading on leg muscle oxygenation and blood volume during high-intensity exercise in chronic heart failure. Am J Physiol Heart Circ Physiol. 2008 Jun;294(6):H2465-72. doi: 10.1152/ajpheart.91520.2007. Epub 2008 Mar 28. PMID 18375714
- [Background] Oliveira MF, Rodrigues MK, Treptow E, Cunha TM, Ferreira EM, Neder JA. Effects of oxygen supplementation on cerebral oxygenation during exercise in chronic obstructive pulmonary disease patients not entitled to long-term oxygen therapy. Clin Physiol Funct Imaging. 2012 Jan;32(1):52-8. doi: 10.1111/j.1475-097X.2011.01054.x. Epub 2011 Oct 3. PMID 22152079